CLINICAL TRIAL: NCT03011606
Title: Robotic Surgery After Focal Ablation Therapy
Acronym: RAFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9211QM
Record Dates: First submitted 2015-07-28; First posted 2017-01-05 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Prostate Cancer
Keywords: prostate; ablation; focal; cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Robotic Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Robotic surgery (Experimental): Single arm. All Registered patients will undergo robotic surgery
  Interventions: Procedure: Robotic Surgery

INTERVENTIONS:
Procedure: Robotic Surgery — Robotic Surgery after Focal Ablation Therapy

SUMMARY:
The toxicity of traditional prostate cancer therapies including radical surgery and external beam radiation is well known. This has prompted a move towards focal therapy where only the cancerous part of the prostate is treated.

To date, studies have demonstrated very promising outcomes following focal therapy with the majority of men maintaining their urinary and sexual function after therapy.

In a small proportion of men, disease recurs after focal therapy. The optimal treatment for men with recurrent disease after focal therapy is yet to be defined. Patients may undergo further focal therapy to the recurrent disease, undergo radiation therapy, whole-gland therapy using a minimally invasive approach such as High Intensity Focused Ultrasound (HIFU) or cryotherapy. Alternatively patients may undergo radical surgery where the whole prostate is removed.

To date, the side-effects or toxicity of any treatment for recurrent prostate cancer after focal therapy has not been formally studied.

Traditionally, the side effects of surgery and radiation therapy performed in patients that have already undergone previous prostate cancer treatment have been considerable with high rates of urinary incontinence and erectile dysfunction. However, as focal therapy leaves a significant area of the prostate untreated, the investigators believe surgery after focal prostate therapy will be associated with a much lower incidence of urinary and sexual dysfunction.

The aim of the RAFT study is to characterise the side effects of prostate cancer surgery in men that have undergone prior focal ablation therapy. In addition, the investigators wish to perform a number of basic science studies to attempt to better understand why the patient has experienced recurrent prostate cancer after focal therapy.

ELIGIBILITY:
Inclusion criteria:

1. Willingness to provide informed consent
2. Males aged 18 years and over
3. Histological confirmed recurrent/residual adenocarcinoma of the prostate with Gleason score following primary focal prostate cancer ablation therapy. Biopsy must have been performed within 6 months of screening for the study
4. Prior focal ablation therapy using either High Intensity Focused Ultrasound (HIFU), Cryotherapy, brachytherapy, electroporation or Photodynamic therapy
5. Serum Prostate Specific Antigen (PSA) must be below 20
6. Absence of metastatic disease
7. Life expectancy ≥ 10 years
8. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
9. MRI imaging to suggest urinary sphincter has not been incorporated in prior ablation therapy

Exclusion Criteria:

1. Serious co-existing medical illness such as chronic active autoimmune disease (within the last 6 months).
2. Other active malignancy over the last 5 years that has required systemic therapy excluding:

   1. Adjuvant therapy in the curative setting
   2. Non-melanoma skin cancer
   3. superficial transitional cell carcinoma
3. No willingness to comply with the procedural requirements of this protocol
4. Coagulopathy/ Cirrhosis
5. Severe obesity defined as a BMI greater than 45
6. Inability to tolerate general anaesthesia
7. Prior pelvic fracture
8. Extensive tethering of the rectum caused by prior ablation therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2016-02; Primary Completion 2019-10-21 (Actual); Study Completion 2019-10-21 (Actual)

PRIMARY OUTCOMES:
Safety profile of surgery: This will be quantified using the Clavien-Dindo classification of complications (I-V) | Up to 12 months following surgical procedure
Toxicity profile prior to surgery | Prior to surgery (at -6 to 0 weeks screening visit)
  This will be quantified using the Short-form Expanded Prostate Cancer Index Composite (EPIC)-26 performed prior to surgery. Outcome analysis will be performed for the Bowel, urinary and sexual domains of the questionnaire.
Toxicity profile following surgery | Up to 12 months following surgery
  This will be quantified using the Short-form Expanded Prostate Cancer Index Composite (EPIC)-26 performed at 3-monthly intervals for 12 months following surgery. Outcome analysis will be performed for the Bowel, urinary and sexual domains of the questionnaire.

SECONDARY OUTCOMES:
Oncological outcome | Up to 12 months following surgical procedure
  Will be quantified using Biochemical-free survival. Biochemical recurrence after surgery will be defined according to American Urological Association (AUA) guidance e.g. a post-surgical serum Prostate Specific Antigen (PSA) >=0.2 on 2 separate occasions.
Oncological outcome | Up to 12 months following surgical procedure
  Will be quantified using need for androgen-ablation therapy. Androgen ablation therapy will include the commencement of Bicalutamide or Goserelin therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Cathcart, Study Chair — Queen Mary University London
Locations (2):
- United Kingdom (2):
  - Guys and St Thomas' Hospital, London, London
  - University College London Hospital, London

REFERENCES:
- [Derived] Cathcart P, Ribeiro L, Moore C, Ahmed HU, Leslie T, Arya M, Orczyk C, Hindley RG, Cahill F, Prendergast A, Coetzee C, Yogeswaran Y, Tunna K, Sooriakumaran P, Emberton M. Outcomes of the RAFT trial: robotic surgery after focal therapy. BJU Int. 2021 Oct;128(4):504-510. doi: 10.1111/bju.15432. Epub 2021 May 13. PMID 33891378